CLINICAL TRIAL: NCT05387850
Title: Association of Clinical Frailty Assessment With Adverse Postoperative Outcomes and Quality of Life in Elderly Non-cardiac Surgery Patients: a Prospective Study
Brief Title: Clinical Frailty Assessment and Postoperative Adverse Outcomes and Quality of Life in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Xiangya Hospital of Central South University (Other); Beijing Anzhen Hospital (Other); Central South University (Other); Peking University People's Hospital (Other); Zhejiang University (Other); Fudan University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); China-Japan Friendship Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Taihe Hospital (Other); Zhejiang Provincial People's Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-Frailty-001
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Perioperative Complications
Keywords: frailty assessment; non-cardiac surgery; Elderly patients; Adverse outcomes after surgery; Frailty scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients over the age of 65: Elderly patients over the age of 65 undergoing elective non-cardiac surgery
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The frailty index may represent a useful decision support tool to optimize modifiable drivers of the quality and cost of digestive surgery care. However, classical indices are cumbersome to compute and often require unavailable data. The number of operations in the elderly is gradually increasing, and the prevention and treatment of adverse postoperative outcomes has become the focus of clinical attention. More recently, clinicians have focused more on the association between frailty and adverse postoperative outcomes, but this has not been rigorously applied to long-term prospective studies in older patients.

DETAILED DESCRIPTION:
As the population aging is speeding up, senile diseases have become a significant and severe public health problem, influencing national health. More than 20 million elderly patients undergo surgery each year in China, accounting for a quarter of the population who undergo surgery. Advanced age and comorbid diseases render the elderly at increased risk of postoperative morbidity and mortality. The incidence of postoperative complications is twice as non-elderly patients, and mortality rates are five times higher than non elderly patients. Thus, it is a significant challenge to safely and stably ensure the elderly in an optimal perioperative period.

Elderly patients continue to pose a major threat to the world's rapidly ageing population due to high rates of surgery and postoperative complications in elderly patients. Therefore, optimizing perioperative management strategies for elderly patients remains one of the biggest challenges facing clinicians.

Frailty is a multidimensional clinical syndrome characterized by vulnerability to dependence and increased mortality when exposed to stressors. It is often clinically described as a lack of physiological reserve, manifested as a loss of physical ability, metabolic function, and cognitive abilities. A systematic review of studies of patients in general surgery reported that the prevalence of prefrailty was estimated to be between 11.3% and 45.8%, while the prevalence of frailty was estimated to be between 10.4% and 37.0%.

Although clinicians or relatives may be aware of frailty, there is currently no standardized clinical gold-standard assessment tool to widely use and quantify frailty.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric surgical patients ≥65 years old
* non-selective cardiac surgery

Exclusion Criteria:

* Missing or incomplete patient follow-up records
* ASA degree V
* Delirium before surgery
* Patient refused to enroll

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: hospital based group
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
mortality | up to 1 month
  postoperative all-cause mortality

SECONDARY OUTCOMES:
the incidence of postoperative delirium | During hospitalization (up to 1 month)
  the incidence of postoperative delirium (3D-CAM scale).Delirium was defined as acute, transient, fluctuating, and usually reversible disturbances in attention, cognition, or attention level. It was assessed every 12 hours by trained nurses using the confusion assessment method (CAM).
postoperative sleep quality | 6 months after surgery
  The PSQI measures sleep quality retrospectively over the previous month using self-report/recall; it consists of nineteen individual items which evaluate the seven components of sleep quality: (1) sleep duration; (2) sleep disturbance; (3) sleep latency; (4) daytime dysfunction due to sleepiness; (5) sleep efficiency; (6) overall sleep quality; and (7) sleep medication usageThese seven component scores (scored 0-3) are added together to yield one global score between 0-21, with higher scores indicating worse sleep quality . A global PSQI score ≤5 indicates good sleep quality and >5 indicates poor sleep quality.
anxiety state and postoperative depression state | 12 months
  The GAD-7 asks how often people have suffered from the seven core symptoms of GAD within the last two weeks with the response options being 'not at all', 'on some days', 'on more than half of the days' and 'almost every day' (scored 0-3, with a total score ranging from 0 to 21) . The GAD-7 has been validated within a large sample of patients in a primary care setting, and within a large general population sample in Germany.The higher the score, the worse the situation.
postoperative quality of life evaluation | 12 months
  Patients'quality of life was assessed through telephone interviews 12 months after surgery using the EQ5D. EQ5D is a measure of health status, assessing daily activities, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension consists of a 3-level response: no problems, moderate problems, or severe problems. A scoring algorithm is available by which each health status description can be expressed as an overall score using the published Chinese tariffs for the Chinese population,12 ranging from 0 (death) to 1 (full health). EQ5Dquestionnaires were acquired according to the script for telephone administration of the EQ5D5L simplified Chinese version for China through telephone interviews 12 months after surgery.
postoperative depression state (PHQ-9) Scale) | 12 months
  Primary outcomes were depression (Patient Health Questionnaire 9 (PHQ-9)).Depression was evaluated using the Chinese version of the patient health questionnaire (PHQ-9), which has nine items measuring self-assessed depressive symptoms experienced during the previous 2 weeks. It uses a 4-point Likert-type scale (0 = never, 1 = sometimes, 2 = more than once a week, and 3 = almost every day). The total score ranges from 0 to 27, and higher scores indicate more depressive symptoms. Scores of 10 and 15 represent cutpoints for moderate and moderately severe depression, respectively. The Chinese version of the PHQ-9 has shown good psychometric properties with reported Cronbach's α of 0.86.
adverse postoperative outcomes | up to 1 month
  Postoperative adverse outcomes include stroke, delirium, major adverse cardiac events, pneumonia, infection, acute renal failure, etc

CONTACTS AND LOCATIONS:
Overall Officials: Mi Weidong, PhD, Study Chair — Chinese PLA hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided